CLINICAL TRIAL: NCT04605809
Title: Effects of Combined Motor and Cognitive Training on Physical Fitness and Brain Fitness in Pre-frail Elderly
Brief Title: Effects of Combined Motor and Cognitive Training in Pre-frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Li-Ling Chuang, Associated Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST 109-2314-B-182-030
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pre-frail Elderly
Keywords: pre-frail, physical fitness, brain fitness, dual-task
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- combined motor and cognitive training (Experimental): The combined motor and cognitive training group will undertake physical fitness training under sitting and standing, walking training while sequentially or simultaneously perform cognitive training.
  Interventions: Device: combined motor and cognitive training
- motor training alone (Active Comparator): The motor training alone group will train the same set of physical fitness training while sitting, standing, and walking as the combined motor and cognitive training group.
  Interventions: Device: motor training alone
- cognitive training alone (Active Comparator): The cognitive training alone group will train the same set of cognitive training while sitting as the combined motor and cognitive training group.
  Interventions: Device: cognitive training alone
- no intervention control group. (No Intervention): No intervention control group will maintain habit and daily activity.

INTERVENTIONS:
Device: combined motor and cognitive training — The combined motor and cognitive training group will receive physical fitness training under sitting and standing, walking training while sequentially or simultaneously perform cognitive training for 45 minutes per session, 3 times a week for 4 weeks.
  Arms: combined motor and cognitive training
Device: motor training alone — The motor training alone group will receive the same set of physical fitness training while sitting, standing, and walking as the combined motor and cognitive training group for 45 minutes per session, 3 times a week for 4 weeks.
  Arms: motor training alone
Device: cognitive training alone — The cognitive training alone group will receive the same set of cognitive training while sitting as the combined motor and cognitive training group for 45 minutes per session, 3 times a week for 4 weeks.
  Arms: cognitive training alone

SUMMARY:
The objective of this study is to investigate psychometric properties of dual-task walking assessments and compare effects of combined motor and cognitive training on physical fitness, brain fitness, and dual-task walking performance in pre-frail elderly. Specifically, we will investigate psychometric properties (i.e. reliability and validity) of dual-task walking assessments for pre-frail elderly (Aim 1). The second aim of this study is to compare the effects of combined motor and cognitive training vs. motor training alone vs. cognitive training alone vs. no intervention control on physical fitness, brain fitness, and dual-task walking performance in pre-frail elderly (Aim 2). The third aim of this study is to elucidate the effects of combined motor and cognitive training on patterns of cognitive motor interference in pre-frail elderly (Aim 3).

DETAILED DESCRIPTION:
A metric analysis and comparative efficacy research will be conducted. Eighty-four pre-frail elderly will receive dual-task walking assessments twice at pretreatment with a 1-week interval for test-retest assessment and investigation of the reliability and validity of outcome measures. The primary outcome measure of the dual-task walking assessments will include walking at preferred speed and fast speed and simultaneously perform serial three subtractions and the Stroop task. Concurrent validity will be studied to validate the dual-task walking measures with each other and with the item 14 of the mini-Balance Evaluation Systems test (Mini-BESTest), dual-task Timed-up-and-Go test (dual-TUG), and 6-min walk test obtain concurrently for assessing dual-task ability. A comparative efficacy research is a single-blind, randomized controlled trial, which will be conducted at medical centers. Pre-frail elderly will be randomized to combined motor and cognitive training, motor training alone, cognitive training alone, or no intervention control group. All three training groups will receive interventions 3 times a week for 4 weeks. The combined motor and cognitive training group will undertake physical fitness training under sitting and standing, walking training while sequentially or simultaneously perform cognitive training. The motor training alone group will train the same set of physical fitness training while sitting, standing, and walking as the combined motor and cognitive training group. The cognitive training alone group will train the same set of cognitive training while sitting as the combined motor and cognitive training group. No intervention control group will maintain habit and daily activity. A blinded assessor will administer three assessments. All participants will be examined physical fitness and brain fitness at baseline twice, and post intervention. The primary outcome measures will be components of physical fitness (cardiopulmonary fitness, muscle fitness, flexibility, body composition, and balance)and brain fitness (information processing speed, working memory, response inhibition, spatial memory, and selective attention). The secondary outcome measures will be gait and cognitive performance under dual-task conditions, dual-Timed Up and Go test, the Mini-BESTest, Functional Gait Assessment, and 6-minute Walk Test, Repeated measure ANOVA will be used to compare measurements at baseline and after training among the groups.

ELIGIBILITY:
Inclusion Criteria:

* age more than 65 years old
* fit one of the criteria for pre-frail definition: (1) body weight lost more than 3 kg or 5% as compared to last year; (2) unable to compete 5 times of Sit to Stand test within 15 seconds; (3 ) more than 3 days fatigue feeling or lack of motivation doing things.
* able to walk 10 meters
* no severe vision, hearing, cognition, and language problems.
* understand instruction (MoCA score>26)

Exclusion Criteria:

* neurological or musculoskeletal diagnosis that affects walking
* cognitive impairment (MoCA<26)
* unable to stand for at least 2 minutes
* moderate to severe high blood pressure (systolic blood pressure more than 160 mmHg and diastolic blood pressure more than 100 mmHg)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 1 minute
  weight and height will be combined to report BMI in kg/m^2 measure body composition.
Waist to hip ratio | 1 minute
  waist to hip ratio measure body composition.
2-Minute Step Test | 2 minutes
  This test measures aerobic endurance. It requires the subjects march in place as fast as possible for 2 minutes while lifting the knees to a height midway between their patella and iliac crests while standing. The score is the number of right-knee reaches the required height completed in 2 minutes.
Chair Stand and Reach Test | 1 minutes
  This test measures lower body flexibility, especially hamstrings. The subject sits on the edge of a chair (placed against a wall for safety). One foot must remain flat on the floor. The other leg is extended forward with the knee straight, heel on the floot, and ankle bent at 90 degree. Place one hand on the top of the other with tips of the middle fingers even. Instruct the subject to inhale, and then as the exhale, reach forward toward the toes by bending at the hip. Knee the back straight and head up. Avoid bouncing or quick movements, and pain. Keep the knee straight , and hold the reach for 2 seconds. The distance is measured between the tip of the fingertips and the toes. If the fingertips touch toes then the score is zero. If they do not touch, measure the distance between the fingers and the toes as a negative score. If they overlap, measure by how much of the distance as a positive score.
Back Scratch Test | 1 minutes
  This test measures upper body flexibility, especially shoulder movement. This test requires the subject in standing position. Place one hand behind the head and back over the shoulder, and reach as far as possible down the middle of his/her back, his/her psalm touching his/her body and the fingers directed downwards. Place the other arm behind his/her back, palsm facing outward and fingers upward and reach up as far as possible attempting to touch or overlap the middle fingers of both hands. The examiner measures the distance between the tips of the middle fingers. If the fingertips touch, the score is zero. If they do not touch, measure the distance between the fingertips as a negative score. If they overlap, measure by how much of the distance as a positive score.
Arm Curl Test | 1 minutes
  This test measures upper body strength and endurance. The subject sits on a chair, holding the weight in the hand using a suitcase grip (palm facing towards the body) with the arm in a vertically down position beside the chair. Brace the upper arm against the body so that only the lower arm is moving (the examiner assists to hold the upper arm steady). Curl the arm up through a full range of motion, gradually turning the palm up (flexion with supination). As the arm is lowered through the full range of motion, gradually return to the starting position. The arm must be fully bent and then fully straightened at the elbow. Repeat this action as many times as possible within 30 seconds. The score is the numbers of the dominant arm curl within 30 seconds.
Chair Stand Test | 1 minutes
  This test measures leg strength and endurance. The subject is seated in the middle of the chair, back straight, feet approximately a shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and help against the chest. Have the subject complete as many full stands as possible within 30 seconds. The subject is instructed to fully sit between each stand. The score is the total number of stands within 30 seconds (more than halfway up at the end of 30 seconds counts as a full stand).
8-Foot Up and Go Test | 1 minutes
  This test measures mobility, balance, walking ability, and fall risk in older adults. The subject sits in the chair with his/her back against the chair back. On the command" Go" the subject rises from the chair, walk 2.44 meters at a fast and safe speed, turns, walk back to the chair and sit down. Timing begins at the instruction "Go" and stops when the subject is seated.
One-leg Standing Test | 1 minutes
  This test measures static balance control and is performed with eyes open (focus on an object about 3 feet in front of the subject), arms on the hips. The subject must stand unassisted on one leg and is timed in seconds from the time one foot is flexed off the floor to the time when it touches the ground or the standing leg ot an arm leaves the hips.
Simple Reaction Time Task (SRT) | 1 minute
  It measures information processing speed.In a sitting position, participants will hear a sequential 5 low pitch (500Hz) that are played by a custom-written MatLab program and present stimuli through a wireless headphone. Participants are instructed to respond verbally the pitch of the sound (low) as quickly and as accurately as possible. Before actual measurements, a series of ten auditory stimuli will be practiced. The number of correct responses and reaction time of correct responses provided within testing will be calculated
Serial three subtraction task | 1 minute
  It measures working memory. In this task targeting working memory, participant will be instructed to count backwards by 3s from a two-digit number (eg, subtract 3 from 99 five times as fast as you can). After 2 trials of practice, another 2 trials will be conducted using 2 new number sets. In addition to accuracy and reaction time, the number of correct responses within the given time period of each trial will be calculated.
Stroop task | 1 minute
  It measures response inhibition.The assessment involves showing the participants words written using inks of various colors, and having the participants state the color of the ink. Participants will be asked to name the color with which a color word will be printed, for instance, if the word "blue" is printed in "red" ink, the participant will need to respond "red" to be correct. The words will be displayed on computer screen in front of participants. Participants will be instructed to name colors of a set of words as accurately and as fast as possible. Before actual measurements, a series of five Stroop stimuli will be practiced. The number of correct responses and reaction time of correct responses provided within testing will be recorded. To account for possible speed-accuracy trade-off, a composite score will be calculated by dividing accuracy (% correct responses) by verbal reaction time to indicate cognitive performance.
Auditory Stroop task | 1 minute
  The Auditory Stroop task measures response inhibition (executive function).Inhibitory assessment of auditory Stroop task will include ignoring the distracter stimuli. Participants hear the words "papa" and "mama," spoken in either a male voice or a female voice; participants are instructed to report the voice of the word (papa/mama) as quickly and as accurately as possible, ignoring the actual word presented.
Spatial Memory Task (SM) | 1 minute
  The SM measures spatial memory. A visuospatial cognition task will consist of visualizing and reciting directions. Two visual yellow stimuli on a 3 by 3 grid will be sequentially presented approximately 0.5 second each and then faded. Then participants have to identify the location of the two stimuli and respond verbally the corresponding numbers on a 3 by 3 grid based on the positions.
Choice Reaction Time Task (CRT) | 1 minute
  The CRT measures selective attention. Participants hear either a high pitch (2500 Hz) or a low pitch (500 Hz) and are instructed to verbal report the pitch of the sound (high or low).

SECONDARY OUTCOMES:
gait and cognitive performance under dual-task conditions | 20 minutes
  Participants will walk 10 meters at their preferred speed and at fast speed. A 12-meter walkway will be used for walking testing. In oder to allow the participants to have enough distance to accelerate and decelerate, only the time taken to walk in the middle 10 meters will be recorded by a stopwatch or Physilog sensors (Gait up, Switzerland). The primary gait parameter is gait speed (cm/sec) under dual-task walking conditions using the 10 Meter Walking Test plus the Stroop task. For walking while performing the Stroop task, we will calculate the composite score for the Stroop task under dual-task walking condition by dividing the accuracy (% correct responses) with the reaction time of correct answers (milliseconds) which accounts for speed-accuracy tradeoffs.
dual-task Timed Up and GoTest (dual-TUG Test) | 2 minutes
  The dual-TUG Test is to perform the TUG Test under dual-task conditions (tray carrying and counting backward by 3s). Participants will be asked to perform the TUG test while carrying a tray with glasses (dual-TUG manual) or counting backward by 3s (dual-TUG cognition). The instruction for dual-TUG tests is to walk with your comfortable speed and concurrently perform a secondary task (carry the tray in front of you with both hands without dropping glasses on the tray or counting backward by 3s). The TUG test is often used as an index of dynamic balance of the elderly. At the signal, participants stand up, walk 3 meter, turn, walk back, and sit down again. The score is the time to complete the test measured using a stopwatch.
Mini-Balance Evaluation System Test (Mini-BEST Test) | 10 minutes
  The Mini-BEST test consists of 14 items and includes four subscales: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each item is rated on a three-point ordinal scale (0=severe, 1=moderate, and 2=normal), with a maximum score of 28 points.
Functional Gait Assessment (FGA) | 10 minutes
  The FGA is comprised of 10-item that contains 7 of 8 items (except walking around obstacles) from the Dynamic Gait Index and 3 additional tasks, including walking with a narrow base of support, walking with the eyes closed, and walking backward. Subjects' perfromance of each test item was rated on a 4-point scale (0-3), with the total score ranging between 0 and 30.
6-minute Walk Test | 6 minutes
  Participants walk for 6-minute at comfortable speed to examine their walking endurance.

CONTACTS AND LOCATIONS:
Overall Officials: LLi-Ling Chuang, Ph.D., Principal Investigator — Chang Gung University
Locations (1):
- Mackay Memory Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No